CLINICAL TRIAL: NCT06242964
Title: The Promoting Resilience in Stress Management-Social Needs (PRISM-SN) Intervention for Adolescents and Young Adults With Cancer: A Randomized Controlled Trial
Brief Title: The PRISM-Social Needs (PRISM-SN) Intervention for Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004509
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Social Functioning; Psychosocial Functioning; Coping Skills
MeSH Terms: conditions — Neoplasms; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM-SN Intervention (Experimental): Skill-based psychosocial program
  Interventions: Behavioral: Promoting Resilience in Stress Management - Social Needs (PRISM-SN)
- Usual Care (No Intervention): Standard psychosocial care

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management - Social Needs (PRISM-SN) — The Promoting Resilience in Stress Management - Social Needs (PRISM-SN) intervention is a brief, skill-based psychosocial program. Five core sessions are delivered one-on-one, 1-2 weeks apart, in-person or via videoconference. Sessions teach evidence-based behavioral skills for managing stress, setting goals, reframing negative thoughts, meaning-making, and connecting with others. Each session lasts <60 minutes and is supported by paper-and-pencil or mobile app-based worksheet(s) for learning and practice. A final review session may be completed individually or with a family member, caregiver, or significant other.
  Arms: PRISM-SN Intervention

SUMMARY:
The goal of this study is to establish feasibility, acceptability, and proof-of-concept of an psychosocial intervention adapted to address social health needs of adolescents and young adults (AYAs) newly diagnosed with cancer. The aims of this study are to:

1. Determine if the Promoting Resilience in Stress Management - Social Needs (PRISM-SN) adapted intervention is feasible and acceptable, defined via program uptake and retention and patient-reported feedback.
2. Explore whether PRISM-SN improves social outcomes at 12-week follow-up compared to usual care.

Participants will be randomized to receive usual psychosocial care or the PRISM-SN program. Participants on both arms will complete patient-reported outcome surveys at enrollment and 12-weeks later. Researchers will compare participants who received the PRISM-SN program to those who received usual care to see if the program improves psychosocial outcomes.

DETAILED DESCRIPTION:
In this randomized controlled trial, AYAs newly diagnosed with cancer will be recruited from two sites and randomly assigned to receive usual care alone or usual care with the Promoting Resilience in Stress Management - Social Needs (PRISM-SN) adapted program. PRISM-SN is a skill-based behavioral program that includes 4 core modules plus a newly developed social health module. Participants on both arms with complete a standardized patient-reported outcome survey assessing aspects of social and psychological functioning at enrollment and 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-25 years
* Diagnosed with new malignancy treated with chemotherapy and/or radiation <6-months
* Able to speak in the English language
* Able to read in the English language
* Cognitively able to participate in intervention sessions and complete surveys

Exclusion Criteria:

* Aged <12 or >25 years
* Diagnosed with recurrent malignancy
* Diagnosed with new malignancy >6 months
* Not receiving chemotherapy and/or radiation
* Not able to speak in the English language
* Not able to read in the English language
* Not cognitively able to participate in intervention session or complete surveys

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cancer Behavior Inventory - Social Relationship Coping Efficacy (CBI-SCRE) Measure | 12-weeks
  The Cancer Behavior Inventory - Social Relationship Coping Efficacy measure assesses one's confidence to engage in behaviors that maintain or enhance close social relationships in the context of illness. Ten items are rated 1-10; items are summed, with higher scores reflecting higher social relationship coping efficacy.

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support (MSPSS) | 12-weeks
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a brief tool designed to measure support from family, friends, and a significant other. It includes 12 items with 4 per subscale. Items are rated on a 7-point Likert scale from 1 (very strongly disagree) to 7 (very strongly agree). It has been validated in both adolescents and adults. Mean scale scores ranging from 1-2.9 can be considered low support; 3-5 considered moderate support; and 5.1-7 considered high support.
Snyder Hope Scale | 12-weeks
  The Snyder Hope Scale contains 8 hope items plus 4 filler questions, and measures the overall perception that one's goals can be met. Each item is scored on an 8-point Likert scale; higher scores imply greater levels of hopeful thought patterns.
Patient Reported Outcome Measurement Information System (PROMIS) Pediatric Profile-25 and Family Relationships Subscale | 12-weeks
  The Pediatric Profile-25 (v2.0) includes 25 items assessing health status across 7 domains: physical function mobility, anxiety, depressive symptoms, fatigue, peer relationships, pain interference, and pain intensity. For this study, we will also include the 4-items pediatric family relationships short-form subscale (v1.0). All items are scored on a 5-point Likert scale except for a single pain intensity item scored on a 10-point scale; higher scores indicate more of each domain. Total raw scores are converted to standardized T-scores with a population mean of 50 and a standard deviation of 10.
Connor-Davidson Resilience Scale (CS-RISC) | 12-weeks
  The Connor-Davidson Resilience Scale (CS-RISC) is a reliable and widely used instrument assessing self-perceived resilience. Scores range from 0-40, with higher scores indicating higher self-perceived resilience.
Hospital Anxiety and Depression Scale (HADS) | 12-weeks
  The Hospital Anxiety and Depression Scale (HADS) assesses mixed affective symptoms in patients with serious illness. The scale includes 7 questions for anxiety and 7 for depression. Each is scored from 0-3 for a total range of 0-21 for each subscale. Clinically relevant symptoms are defined as scores of 8 or higher for both anxiety and depression.

OTHER OUTCOMES:
Acceptability of Intervention Measure (AIM) | 12-weeks
  The Acceptability of Intervention Measure (AIM) assess perceived intervention acceptability. It includes 4-items such as "[program] meets my approval," scored 1-5, with higher scores reflecting more acceptability. Scores are averaged across items. This measure will be completed by experimental arm participants only.

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlyn M Fladeboe, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data may be shared upon request. Investigators interested in conducting additional analyses must request data directly from the PI via written correspondence and obtain and provide verification of institutional review board approval.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared after publication of study findings; coded banked data will be available indefinitely.
Access Criteria: Written request to the PI.

REFERENCES:
- [Derived] Fladeboe KM, Fredman G, Maurer SH, Zhou C, Bradford MC, Yi-Frazier JP, Salsman JM, Baker KS, Mack MC, Taylor MR, Rosenberg AR. Feasibility and proof-of-concept of a combined resilience and social connection intervention for adolescents and young adults with cancer: a pilot randomized trial protocol. Pilot Feasibility Stud. 2026 Jan 29. doi: 10.1186/s40814-026-01775-0. Online ahead of print. PMID 41612517